CLINICAL TRIAL: NCT05836428
Title: Biomarker Analysis in COVID and Post-COVID Patients
Brief Title: Biomarker Analysis in Post-COVID Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Laura de Boni, Principal investigator, University Hospital, Bonn
Other Study IDs: 2
Record Dates: First submitted 2023-04-26; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Post-COVID-19 Syndrome
Keywords: persistent headache
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Persistent post-COVID-19 headache: post-COVID-19 patients with persistent headache
  Interventions: Other: no intervention
- controls: Mild Neuro-COVID-19 patients without persistent headache and other neurological diseases
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Headache is one of the most common neurological manifestations of COVID-19. However, it is unclear whether chronic headache after the initial diagnosis, is associated with ongoing damage of the central nervous system. We investigate cpost-COVID-19 patients with persistent headache lasting longer than 3 weeks, to hospitalized acute COVID-19 patients with neurological symptoms and to other non-COVID-19 disease-controls. Readout are neurologial and glial biomarkers in CSF.

DETAILED DESCRIPTION:
Measurements of neuronal and glial markers in CSF were performed on a SIMOA analyzer (Quanterix) using the Neurology 4-Plex A (Nf-L, Tau, GFAP, UCH-L1) kit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COVID, Parkinson's disease, primary headache, Multiples Sclerosis, facial paralysis
* Persistent post-COVID-19 headache after 3 months of infection
* Post COVID-patients without persistent headache
* must be able to perform lumbar puncture

Exclusion criteria

* unknown history of COVID infection
* lumbar puncture not possible

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Biomarker analysis in CSF | after 3 months of initial infection
  Levels of Nf-L, Tau, GFAP, UCH-L1 in CSF

CONTACTS AND LOCATIONS:
Overall Officials: Laura de Boni, MD, Principal Investigator — DLR German Aerospace Center
Locations (1):
- Laura de Boni, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No